CLINICAL TRIAL: NCT05581017
Title: Association of Cephalosporin Resistance in Intraoperative Biliary Cultures with Surgical Site Infections in Patients Undergoing Pancreaticoduodenectomy - a Retrospective Cohort Study
Brief Title: Association of Cephalosporin Resistance and Surgical Site Infections in Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Timo Tarvainen, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: HUS-115-2020-56
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2022-10

CONDITIONS: Surgical Site Infection; Pancreaticoduodenectomy; Biliary Tract Infection Bacterial
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- No PBD: Patients without preoperative biliary drainage before pancreaticoduodenectomy
- PBD < 2 months: Patients who had undergone preoperative biliary drainage and the pancreaticoduodenectomy was in 2 months after the drainage.
  Interventions: Procedure: Preoperative biliary drainage
- PBD ≥ 2 months: Patients who had undergone preoperative biliary drainage and the pancreaticoduodenectomy was at 2 months or later after the drainage.
  Interventions: Procedure: Preoperative biliary drainage

INTERVENTIONS:
Procedure: Preoperative biliary drainage — Preoperative biliary drainage before pancreaticoduodenectomy. Might be needed if the biliary tract in obstructed and the surgery cannot be scheduled in near future.
  Groups: PBD < 2 months; PBD ≥ 2 months

SUMMARY:
Preoperative biliary drainage predisposes the bile to be contaminated with bacteria of the duodenum. These bacteria colonizing the bile are a potential source for surgical site infections after pancreaticoduodenectomy and many international guidelines recommend the use of cephalosporines as microbial prophylaxis before surgery. The aim of this study was to assess the incidence of bacteria in bile, their resistance profiles and association to surgical site infections in relation to timing of surgery after preoperative biliary drainage in order to better guide antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pancreaticoduodenectomy between May 23rd 2016 to October 29th 2020

Exclusion Criteria:

* Patients without intraoperative biliary culture
* Patients with unknown date of preoperative biliary culture

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing pancreaticoduodenectomy in a single high volume center between May 23rd 2016 to October 29th 2020.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Rate of surgical site infections | 30 days post operatively
Prevalence of cephalosporin resistance in intraoperative biliary cultures | At the time of operation

CONTACTS AND LOCATIONS:
Overall Officials: Timo O Tarvainen, MD, Principal Investigator — Gastroenterological Surgery, Helsinki University Hospital
Locations (1):
- Helsinki Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No